CLINICAL TRIAL: NCT04535778
Title: Pilot RCT for COMPASS: an Online CBT Program Treating Anxiety and Low Mood in Long-term Conditions During the COVID-19 Pandemic.
Brief Title: COMPASS Study: an Online Cognitive-behavioural Therapy (CBT) Program Treating Anxiety and Low Mood in Long-term Conditions During the COVID-19 Pandemic
Acronym: COMPASS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: National Multiple Sclerosis Society (Other); Psoriasis Association (Unknown); Crohn's & Colitis UK (Unknown); Kidney Care UK (Other); Shift.ms (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20347
Record Dates: First submitted 2020-08-12; First posted 2020-09-02 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-02

CONDITIONS: Treatment of Illness-related Distress in Physical LTCs

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- COMPASS (Experimental): Participants will be treated with an online CBT program that is specifically tailored to illness-related distress in the context of long-term conditions. Participants will also have access to the standard charity resources.
  Interventions: Behavioral: COMPASS
- Standard charity resources (Active Comparator): Participants will be directed to the standard resources provided by the charities involved in the study.
  Interventions: Behavioral: Standard charity resources

INTERVENTIONS:
Behavioral: COMPASS — An 11 module, therapist-supported online CBT program.
  Arms: COMPASS
Behavioral: Standard charity resources — Resources provided by the charities involved, including supportive listening, online support groups, information resources and local community support groups.
  Arms: Standard charity resources

SUMMARY:
This study is a single-centre, interventional randomised controlled trial.

Participants will be individually randomised to receive either COMPASS online CBT + "usual care" (standard LTC charity support), or usual care only. Randomisation will be stratified by recruiting charity site to ensure a balance of participants with different LTCs across the intervention and control arm. Randomisation will occur using a 1:1 allocation ratio managed by RECAP software.

Participants randomised to COMPASS will receive access to the online program. It consists of 11 online modules which target challenges associated with living with LTC(s) and includes, amongst other things, psycho-education, patient examples, interactive tasks and goal setting. Participants are linked to a therapist; 'guide', who will provide 6 x 30 minute support sessions delivered fortnightly in the format preferred by the client (phone and/or in-site message).

Participants allocated to the usual care control arm will receive the usual care that is available to them via their charity. All charities include a helpline which can be accessed via telephone or email. The helplines at all charities offer one-off emotional and/or informational support provided by people trained in active listening and/or counselling skills. Additional support avenues that can be accessed may include online support groups, local community support groups and informational resources.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 or over
* Have responded to sign posting advise from the LTC charity or responded to an advert placed on a LTC charity website expressing their interest in taking part in the study.
* Speak English to a sufficiently high standard to allow them to interact with digital CBT programs.
* Live in the UK and can provide contact details of their registered general practitioner
* Have an email address to allow them to register with a digital CBT program and have a basic understanding of the internet.
* Scores ≥3 on the shortened patient health questionnaire (PHQ-4) self-report measure of depression and anxiety in relation to their LTC and/or the COVID-19 pandemic.

Exclusion Criteria:

* Evidence of alcohol and/or drug dependency, cognitive impairment, severe mental health disorders, including bipolar disorder or psychosis
* Acute suicidal risk requiring a level of support that cannot be provided by therapists who are supporting patients remotely in their use of digital health interventions.
* Receiving active psychological treatment. Active psychological treatment is defined as receiving treatment from a psychologist/counselor/therapist or engaging with other online psychological treatment interventions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2020-11-16 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Patient Health Questionnaire Anxiety and Depression Scale (PHQ-ADS) | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  A composite measure of Generalised Anxiety Disorder questionnaire (GAD-7) and Patient Health Questionnaire (PHQ-9). Min score = 0, Max score = 48, with higher scores indicating higher levels of distress.

SECONDARY OUTCOMES:
Change in Work and social adjustment scale (WSAS) | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Social functioning. Min score = 0, Max score = 40 , with higher scores indicating greater functional impairment.
Change in EQ-5D-3L | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Quality of life. Min score = 5, Max score = 15 , with higher scores more problems in the scale dimensions.
Change in Illness perception questionnaire - revised (IPQ-R), emotional subscale | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  IPQ-R tailored to COVID-19 to establish emotional responses regarding the COVID-19 pandemic. Min score = 0, Max score = 24 , with higher scores indicating higher emotional responses.
Change in Patient Health Questionnaire - (PHQ-9) | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Depression. Min score = 0, Max score = 27, with higher scores indicating greater depression
Change in Generalised Anxiety Disorder scale (GAD-7) | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Anxiety. Min score = 0, Max score = 21, with higher scores indicating greater anxiety
Change in bespoke illness-related distress measure (2 items) | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Illness-related distress. Developed by research team. Min score = 0, Max score = 6, with higher scores indicating greater distress.
Change in Patient Activation Measure (PAM) short version (13 items). | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Assess knowledge and confidence in illness self-management. Min score = 0, max score = 100, with higher scores indicating greater levels of knowledge and confidence.
The Patient Global Impression Scales of Severity (PGI-S) | At baseline, 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Perceived symptom severity. 1 item. Min = 0, Max = 3, with higher scores indicating greater perceived symptom severity.
The Patient Global Impression Scales of Improvement (PGI-I) | 6 weeks (mid-therapy) and 12 weeks (end of therapy)
  Perceived symptom improvement. 1 item. Min = 0, Max = 6, with higher scores indicating greater perceived symptom deterioration.

CONTACTS AND LOCATIONS:
Overall Officials: Rona Moss-Morris, Principal Investigator — King's College London
Locations (1):
- Health Psychology Section, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The data that support the findings of this study will be available on request from the corresponding author. The data will not be available publicly due to privacy or ethical restrictions.
Supporting Information: CSR
Access Criteria: The data will only be available on request.

REFERENCES:
- [Derived] Picariello F, Hulme K, Seaton N, Hudson JL, Norton S, Wroe A, Moss-Morris R. A randomized controlled trial of a digital cognitive-behavioral therapy program (COMPASS) for managing depression and anxiety related to living with a long-term physical health condition. Psychol Med. 2024 Jun;54(8):1796-1809. doi: 10.1017/S0033291723003756. Epub 2024 Feb 14. PMID 38350600
- [Derived] Hulme K, Hudson JL, Picariello F, Seaton N, Norton S, Wroe A, Moss-Morris R. Clinical efficacy of COMPASS, a digital cognitive-behavioural therapy programme for treating anxiety and depression in patients with long-term physical health conditions: a protocol for randomised controlled trial. BMJ Open. 2021 Oct 25;11(10):e053971. doi: 10.1136/bmjopen-2021-053971. PMID 34697123